CLINICAL TRIAL: NCT02631278
Title: Tissue Effect in Extirpated Uterine Fibroid Tissue Using Existing Olympus Radiofrequency Probes for Fibroids Ablation (Radio Frequency Ablation RFA STUDY )
Brief Title: Radio Frequency Ablation (RFA STUDY )
Acronym: RFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Olympus Winter & Ibe (Unknown)
Responsible Party: Principal Investigator, Prof. Giovanni Scambia, Professor, Catholic University of the Sacred Heart
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 4962/14
Record Dates: First submitted 2015-01-19; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Uterine Myoma
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Other): Intraoperative radiofrequency ablation
  Interventions: Device: Intraoperative radiofrequency ablation

INTERVENTIONS:
Device: Intraoperative radiofrequency ablation — Intra-operative Radiofrequency ablation will be carried out and followed by surgical removal of the treated leiomyoma.
  Other Names: The CelonPower system Olympus

SUMMARY:
The aim of this study is to investigate the safety and feasibility of a radiofrequency (RF) system employing RFITT (CelonProSurge) probes for the ablative treatment of uterine fibroids.

DETAILED DESCRIPTION:
10 consecutive premenopausal women with symptomatic uterine fibroids not responsive to medical therapies (including progestins, oral contraceptives, and anti-inflammatory drugs) will be recruited at our hospital to be submitted to abdominal myomectomy. All patients will be counseled on the potential risks and benefits of the procedure before giving their own written consent.

Procedures will be performed at the hospital and patients will be under general anesthesia.All patients will be submitted to abdominal myomectomy. Target leiomyomas will be intramural, 5-15 cm in diameter. Intra-operative RF ablation will be carried out followed by surgical removal of the treated leiomyoma. After the removing of the fibroid, it will be send to the pathologist. Specimens of fibroid will be fixed immediately in 10% neutral formaline solution for approximately 3h, then embedded in paraffin, cut into 4mm section and stained with along the direction of the RFA electrode. Pathologic confirmation of ablation will be assessed as follows: the specimens of leiomyoma will be examined grossly for the histologic leiomyoma subtype and for pathologic findings representing treatment, including necrosis, hemorrhage, or fibrosis, using hematoxylin and eosin staining. Treated areas will be measured for their largest orthogonal dimensions in the planar cut surface with the third dimension estimated by summing the affected 0.5-cm-thick sagittal planes. RF ablation volumes will be calculated using the prolate ellipsoid formula. The relationship between thermal dose estimates and pathology will be assessed using Bland-Altman analyses and intra-class correlations. The surgical procedure will be concluded as usual with the same steps of standard approach.

ELIGIBILITY:
Inclusion Criteria:

1. premenopausal women, 25 years of age or older;
2. presence of fibroid-related symptoms (menorrhagia, pelvic pain and/or bulk symptoms) not responsive to medical therapy;
3. uteri <20-week gestational size on pelvic examination;
4. one myoma 5-15 cm in diameter as measured by transvaginal ultrasound;
5. desire for uterine preservation;
6. normal coagulation profile;
7. normal Pap test result in the last year,
8. hemoglobin level of 10.0 g/dL or more at the time of treatment.

Exclusion Criteria:

1. pedunculated subserosal or intracavitary myomas,
2. a history of pelvic malignancy,
3. presence of cervical dysplasia,
4. a prior procedure to treat or remove myomas,
5. contraindications to general anesthesia or abdominal surgery.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Estimation termal dose | Intraoperative time
  Specimens of fibroid will be fixed immediately in 10% neutral formaline solution for approximately 3h, then they will be embedded in paraffin, cut into 4mm section and stained with along the direction of the RFA electrode. Pathologic confirmation of ablation will be assessed as follows: the specimens of leiomyoma will be examined grossly for the histologic leiomyoma subtype and for pathologic findings representing treatment, including necrosis, hemorrhage, or fibrosis, using hematoxylin and eosin staining. Treated areas will be measured for their largest orthogonal dimensions in the planar cut surface with the third dimension estimated by summing the affected 0.5-cm-thick sagittal planes. RF ablation volumes will be calculated using the prolate ellipsoid formula. The relationship between thermal dose estimates and pathology will be assessed using Bland-Altman analyses and intra-class correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Scambia, MD, Principal Investigator — Catholic University of Sacred Heart - Rome
Locations (2):
- Italy (2):
  - Catholic University of Sacred Heart Rome,, Rome, Rome
  - Catholic University of Sacred Heart, Rome, Rome

REFERENCES:
- [Background] Bergamini V, Ghezzi F, Cromi A, Bellini G, Zanconato G, Scarperi S, Franchi M. Laparoscopic radiofrequency thermal ablation: a new approach to symptomatic uterine myomas. Am J Obstet Gynecol. 2005 Mar;192(3):768-73. doi: 10.1016/j.ajog.2004.10.591. PMID 15746670
- [Background] Mirza AN, Fornage BD, Sneige N, Kuerer HM, Newman LA, Ames FC, Singletary SE. Radiofrequency ablation of solid tumors. Cancer J. 2001 Mar-Apr;7(2):95-102. PMID 11324771
- [Background] Gazelle GS, Goldberg SN, Solbiati L, Livraghi T. Tumor ablation with radio-frequency energy. Radiology. 2000 Dec;217(3):633-46. doi: 10.1148/radiology.217.3.r00dc26633. PMID 11110923
- [Background] Kawamura K, Suzuki K, Tsugawa R, Taniguchi N, Matsunou H. Influence of RF capacitive heating on the alpha 1-adrenergic receptors of rat prostates. Eur Urol. 1994;25(4):330-3. doi: 10.1159/000475312. PMID 8056027
- [Background] Ichimura T, Kawamura N, Ito F, Shibata S, Minakuchi K, Tsujimura A, Umesaki N, Ogita S. Correlation between the growth of uterine leiomyomata and estrogen and progesterone receptor content in needle biopsy specimens. Fertil Steril. 1998 Nov;70(5):967-71. doi: 10.1016/s0015-0282(98)00300-8. PMID 9806586